CLINICAL TRIAL: NCT00080509
Title: A Phase 2 Study of KOS-862, Administered Intravenously Weekly for 3 Weeks Every 4 Weeks, in Patients With Non-Small Cell Lung Cancer Who Have Progressed Following Initial Therapy for Advanced or Metastatic Disease
Brief Title: Effectiveness of KOS-862 in the Treatment of Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOS-201/NO17352
Record Dates: First submitted 2004-04-05; First posted 2004-04-07 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2009-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — desoxyepothilone B

INTERVENTIONS:
Drug: KOS-862

SUMMARY:
The purpose of this study is to determine whether a potential drug known as KOS-862 or "Epothilone D" has an effect as a 2nd line treatment in non-small cell lung cancer (NSCLC) for patients having failed one prior platinum-containing chemotherapy regimen.

DETAILED DESCRIPTION:
To determine the antitumor activity, based on the confirmed objective response rate, of KOS-862, administered intravenously weekly for 3 weeks every 4 weeks, in patients with non-small cell lung cancer (NSCLC) whose disease has progressed following initial chemotherapy for advanced or metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Measurable disease
* One previous treatment of a platinum based drug such as cisplatin or carboplatin
* At least 3 weeks since last surgery/radiation/chemotherapy

Exclusion Criteria:

* Brain metastases
* Changes in the rhythm of your heart that are considered significant as determined by an ECG tracing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85
Dates: Start 2003-12; Study Completion 2004-11

PRIMARY OUTCOMES:
NSCLC